CLINICAL TRIAL: NCT00304668
Title: A Phase I/II Single-Centre Double-Blinded Randomized Study of the Safety and Tolerability of TMC120 Vaginal Microbicide Gel (TMC120 Gel-002) vs. HEC-Based Universal Placebo Gel in Healthy HIV-Negative Women.
Brief Title: A Safety Study of Dapivirine (TMC120) Vaginal Microbicide Gel in South Africa
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM005A
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2006-05

CONDITIONS: HIV Infections
Keywords: HIV-1; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: dapivirine (TMC120) vaginal gel

SUMMARY:
Approximately 42 HIV-negative women, aged >18 and < 50, will be enrolled in this study. Each volunteer will have a 2:1 chance of receiving Dapivirine Gel-002 versus placebo. The volunteers will receive investigational product for a total of 42 days.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative
* Willing to participate and sign an informed consent form
* Willing to be tested for HIV, use an experimental vaginal gel, and to be randomized to a study group that includes the possibility of being assigned to a placebo group.
* Willing to use two forms of contraception during the study
* Willing to undergo pelvic examinations with colposcopy and photographic documentation according to the protocol throughout the study.
* Have a regular menstrual cycle defined as having a minimum of 21 days and a maximum of 36 days between menses

Exclusion Criteria:

* Currently pregnant or breast-feeding
* Clinically detectable genital abnormality on the vulva, vaginal walls or cervix
* Laboratory confirmed gonorrhea, chlamydia, trichomonas, syphilis, or vaginal candidiasis or clinically diagnosed GUD or active HSV-2 lesion
* Breakthrough bleeding or gynecologic surgery within 60 days prior to randomization
* Symptomatic bacterial vaginosis at Screening and unwilling to undergo treatment.
* Women who require treatment for tuberculosis (TB) within 21 days prior to randomization.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Local and systemic safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Zeda Rosenberg, ScD, Study Director — Beijing Immupeutics Medicine Technology Limited